CLINICAL TRIAL: NCT03713658
Title: A Pilot-Study in Rwandan Health Care Settings to Examine the Feasibility of a Large Pragmatic Clinical Study to Assess the Value of Paliperidone Palmitate in Rwanda
Brief Title: A Study to Evaluate the Ability of Conducting a Study of Oral Risperidone Followed by Paliperidone Palmitate in Rwandan Healthcare Facilities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CR108551; R092670PSY4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Risperidone (Experimental): Participants will receive 3 milligram (mg) oral risperidone tablets once daily for up to one Week to determine tolerability based on investigator review.
  Interventions: Drug: Risperidone 3 mg
- Paliperidone Palmitate Once Monthly (PP1M) (Experimental): Participants will receive 50, 75, 100 or 150 mg eq. ([paliperidone palmitate] mg equivalent [to paliperidone]) long acting formulation of paliperidone palmitate once monthly (PP1M) intramuscular injection for 4 months (17 weeks) plus option to continue 3 more months if not stabilized depending on the participant's clinical safety, tolerability and efficacy requirements.
  Interventions: Drug: Paliperidone Palmitate 50 mg eq.; Drug: Paliperidone Palmitate 75 mg eq.; Drug: Paliperidone Palmitate 100 mg eq.; Drug: Paliperidone Palmitate 150 mg eq.
- Paliperidone Palmitate Every 3 Months (PP3M) (Experimental): Participants will receive 175, 263, 350 or 525 mg eq. ([paliperidone palmitate] mg equivalent [to paliperidone]) long acting formulation of paliperidone palmitate every 3 months (PP3M) intramuscular injection for 24 Weeks.
  Interventions: Drug: Paliperidone Palmitate 175 mg eq.; Drug: Paliperidone Palmitate 263 mg eq.; Drug: Paliperidone Palmitate 350 mg eq.; Drug: Paliperidone Palmitate 525 mg eq.

INTERVENTIONS:
Drug: Risperidone 3 mg — Participants will receive 3 mg oral risperidone tablets once daily for up to one Week.
  Arms: Oral Risperidone
Drug: Paliperidone Palmitate 50 mg eq. — Participants will receive 50 mg eq. PP1M intramuscular injection for 17 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Once Monthly (PP1M)
Drug: Paliperidone Palmitate 75 mg eq. — Participants will receive 75 mg eq. PP1M intramuscular injection for 17 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Once Monthly (PP1M)
Drug: Paliperidone Palmitate 100 mg eq. — Participants will receive 100 mg eq. PP1M intramuscular injection for 17 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Once Monthly (PP1M)
Drug: Paliperidone Palmitate 150 mg eq. — Participants will receive 150 mg eq. PP1M intramuscular injection for 17 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Once Monthly (PP1M)
Drug: Paliperidone Palmitate 175 mg eq. — Participants will receive 175 mg eq. PP3M intramuscular injection for 24 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Every 3 Months (PP3M)
Drug: Paliperidone Palmitate 263 mg eq. — Participants will receive 263 mg eq. PP3M intramuscular injection for 24 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Every 3 Months (PP3M)
Drug: Paliperidone Palmitate 350 mg eq. — Participants will receive 350 mg eq. PP3M intramuscular injection for 24 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Every 3 Months (PP3M)
Drug: Paliperidone Palmitate 525 mg eq. — Participants will receive 525 mg eq. PP3M intramuscular injection for 24 Weeks.
  Other Names: R092670
  Arms: Paliperidone Palmitate Every 3 Months (PP3M)

SUMMARY:
The purpose of this study is to evaluate the feasibility of conducting a study of oral risperidone followed by paliperidone palmitate for once monthly (PP1M) and paliperidone palmitate for every 3 months (PP3M) in rwandan healthcare facilities with mental healthcare capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of schizophrenia by mini international neuropsychiatric interview (MINI)- Screen/ MINI (Module K) that requires treatment initiation or a change in treatment to better address safety or efficacy limitations of current treatment
* Participants at least moderately ill as measured by the clinical global impressions - severity of schizophrenia (CGI-SS) scale for schizophrenia, or experiencing poorly tolerated side effects from their current medications, or having difficulty with adequate adherence to treatment, per the investigator's judgement
* Participants have a primary caregiver who is willing to participate in this study (caregiver should be knowledgeable about the participant's condition and is expected to be with the participant for greater than (>) 24 hours each week for the duration of the study)
* Participants able to give consent to participate in a clinical study that includes treatment with risperidone and long-acting injectable formulations of paliperidone palmitate. Participants must be willing to receive injections. The participant and the caregiver participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Participants must be willing and able to provide responses for all self-administered questionnaires

Exclusion Criteria:

* Participants have a physical, mental, or legal incapacity that prevents a valid consent or capacity to complete about 12 months of treatment with antipsychotic medication and compliance with this study protocol
* Participants with history of organic brain syndromes, comorbid psychiatric and/or physical illnesses, or significant comorbid substance abuse that is likely to interfere with understanding of or compliance with study requirements
* Participants with known allergies, hypersensitivity, or intolerance to risperidone or paliperidone palmitate or their excipients
* Participants with poor prior response to risperidone
* Participants who received an investigational medication (including investigational vaccines) or used an invasive investigational medical device within 30 days before the planned first dose of study medication, or is currently enrolled in an investigational study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Successful Completion of Study Procedures | Up to Week 46
  Percentage of participants with successful completion of study procedures related to diagnosis and outcome measures assessment will be reported.
Percentage of Participants With Successful Delivery of Risperidone/PP1M/PP3M for the Duration of the Study | Up to Week 46
  Percentage of participants with successful delivery of risperidone/PP1M/PP3M for the duration of the study will be reported.
Percentage of Participants With Successful Administration of Risperidone/PP1M/PP3M Throughout the Study | Up to Week 46
  Percentage of participants with successful administration of risperidone/PP1M/PP3M throughout the study will be reported.
Quality of Life as Assessed by World Health Organization Quality of Life Scale Brief Version (WHO QoL-BREF) Total Score | Up to Week 46
  The WHO QoL-BREF is a 25 item scale used to assess the quality of life. All items are rated on a five-point likert scale using response categories such as 1 represents very poor and 5 represents very well with a possible maximum score of 125 and a minimum score of 25.
Clinician Satisfaction as Assessed by Clinician Satisfaction Rating Scale Score | Up to Week 46
  The Clinician Satisfaction Rating is a 4-item scale. Two items use a Likert scale with a six-point range from 0 (definitively not) to 6 (definitely) and two items are multiple-choice (example, "select all that apply"). The scale will be used to assess the acceptability and/or burden for the provider associated with the study including treatment with long-acting injectables (LAIs).

SECONDARY OUTCOMES:
Number of Participants Who Met Mini-International Neuropsychiatric Interview (MINI)-MINI Screen and Module K Criteria | Up to Week 46
  The MINI-Screen is a structured and standardized diagnostic interview used to determine the most common psychiatric disorders according to axis I diagnostic and statistical manual of mental disorders-fourth edition text revision (DSM-IV-TR) and the international classification of diseases and related health problems (ICD-10). The MINI-screen will be administered to participants for preselection by a qualified psychiatric professional. If this step is passed, then Module K of MINI will be applied by a medical doctor (preferably a psychiatrist) or a psychologist in order to confirm the diagnosis of schizophrenia and to determine if there are other psychiatric conditions present. Number of participants who met MINI criteria will be assessed.
Number of Participants Intended to Complete/Attend Next Visit as Assessed by Intent-to-Attend (ITA) Plus Assessment Scale | Up to Week 46
  The ITA-Plus scale is a single Likert scale question with a range of 0 indicates definitely not attending to 6 indicates definitely attending that will be used to estimate the likelihood of completing the study or attending the next visit to provides qualitative feedback on why completion/attendance may not occur. Number of participants intended to complete/attend next visit will be assessed.
Direct Cost Assessment of Schizophrenia Care as Assessed by Client Service Receipt Inventory (CSRI) Scale Score | Up to Week 46
  The CSRI scale will be used to assess the costs of schizophrenia care for participants, caregivers, and health care providers, especially direct costs.
Indirect Cost Assessment of Schizophrenia Care as Assessed by Cost Assessment Questionnaire (CAQ) | Up to Week 46
  The CAQ will be used to assess the costs of schizophrenia care for participants, caregivers, and health care providers, especially indirect costs.
Change From Baseline in Sheehan Disability Scale (SDS) Total Score | Baseline up to Week 46
  SDS will be used to assess the functioning of participants with schizophrenia. It has participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. First three items assess disruption of 1 work/school, 2 social life, 3 family life/home responsibilities using a 0 (no impairment) - 10 (most severe impairment). Score for first 3 items are summed to create total score of 0-30 where higher score indicates greater impairment and a negative change in score indicates improvement.
Number of Participants With Adverse Events (AEs) as a Measure of Safety | Up to Week 46
  Safety will be assessed by AEs along with concomitant medications, past medical history, and demographics of participants who will participate in this study. An adverse event is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the medication. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Psychosis as Assessed by Mental Illness With Lay Evidence (SMILE) Scale Score | Up to Week 46
  The Psychosis module of the SMILE will be used to assess the clinical symptoms of schizophrenia. It is a 15-item Likert scale covering questions to describe participants condition like if they have kept the body neat and clean, difficulty in completing routine tasks, talked to themselves etc with answers on a point range of 0 (Never) to 5 (All the time). It uses 7-day recall period. Both the participant and caregiver participant will complete this scale.
Clinical Global Impression - Severity of Schizophrenia (CGI-SS) Scale Total Score | Up to Week 46
  The CGI-SS will be used to provide a clinical measure of the severity of schizophrenia. It is a single-item Likert scale with a 7-point range (0 indicates none to 7 indicates extreme symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Rwanda (3):
  - CARAES Ndera Neuro-Psychiatric Hospital, Kigali
  - Ruhengeri Referral Hospital, Public Hospital, Musanze District
  - Kibungo Referral Hospital, Ngoma District

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Alphs L, Turkoz I, Smith-Swintosky V, Keenan A, Abraham E, Schotte A, Hooker E, Damascene Iyamuremye J, Kayiteshonga Y, Bizoza R, Mancevski B. Feasibility study to evaluate capabilities for conducting psychiatric clinical research within the Rwandan mental healthcare system. BMJ Open. 2023 Apr 18;13(4):e064675. doi: 10.1136/bmjopen-2022-064675. PMID 37072361
- See also: A Pilot-Study in Rwandan Health Care Settings to Examine the Feasibility of a Large Pragmatic Clinical Study to Assess the Value of Paliperidone Palmitate in Rwanda — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108551&attachmentIdentifier=7d07c1a7-2442-4cfe-8f26-120828a27cd7&fileName=CR108551_CSR_Synopsis.pdf&versionIdentifier=